CLINICAL TRIAL: NCT06419517
Title: Efficacy of PFMT and sEMG-triggered Electrostimulation in Treating the Very Weak Pelvic Floor: a Randomized Clinical Trial
Brief Title: Pelvic Muscle Training and Electrostimulation to Treat Weak Pelvic Floor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Collaborators: BEACMED s.r.l. (Unknown)
Responsible Party: Principal Investigator, DR. GIANFRANCO LAMBERTI, Director, Rehabilitative Medicine Department, Azienda Unita Sanitaria Locale di Piacenza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-0000035
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Pelvic Floor Muscle Weakness; Incontinence Stress; Electricity; Effects; Muscle Weakness Condition
Keywords: Pelvic Floor Muscle Weakness; Electrical Stimulation; Pelvic Floor Muscle Training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Multicentric Prospective Clinical Trial with two parallel arms
Who Masked: Participant, Investigator
Masking Description: Double (participants, principal investigator). To improve the effect of blindness, participants were informed that the trial intended to compare the effects of two Electrical Stimulation (ES) methods for Stress Urinary Incontinence (SUI)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Pelvic Floor Muscle Training + EMG-triggered ES (Experimental): Group A (supervised PFMT + EMG-triggered ES) Supervised Pelvic Floor Muscle Training Twenty sessions will be applied, 2 per week for ten weeks
  Stimulation parameters:
  Duration: 15 min Electrode placement: vaginal probe Frequency: 50 Hz. - Pulse width 250 microseconds Intensity: to motor response (activation of PFM) Number of sessions: 20 Ramp up/down: 1 sec.
  Interventions: Device: EMG-triggered ES; Other: Pelvic Floor Muscle Training
- Supervised PFMT + sham EMG-triggered ES) (Active Comparator): Group B: Supervised PFMT + sham EMG-triggered ES) Supervised Pelvic Floor Muscle Training Twenty sessions will be applied, 2 per week for ten weeks
  Stimulation parameters:
  Duration: 15 min Electrode placement: vaginal probe model xx Frequency: 2 Hz. - Pulse width 10 microseconds Intensity: to sensory response Number of sessions: 20 Ramp up/down: 1 sec.
  Interventions: Other: Pelvic Floor Muscle Training

INTERVENTIONS:
Device: EMG-triggered ES — The ES treatment protocol consisted of daily endovaginal electrostimulation sessions for four weeks. We used a portable unit EVOSTIM ®, which allowed us to use different frequencies and length of impulse and a probe Perisphera ® The average current intensity was adjusted according to the sensation of discomfort in each patient.
  Other Names: Pelvic Floor Muscle Training
  Arms: Supervised Pelvic Floor Muscle Training + EMG-triggered ES
Other: Pelvic Floor Muscle Training — Standardization of the supervised PFMT To achieve standardization of supervised PFMT treatments, a written protocol for the physiotherapeutic examinations and PFMT program will be provided to the physiotherapists (or nurse or midwife) delivering the treatments (See Additional file).
  Other Names: EMG-triggered ES

SUMMARY:
This research will determine 1) whether the very weak pelvic floor can be improved with surface electromyography (s-EMG)-triggered electrostimulation added to pelvic floor muscle training and 2) whether sEMG-triggered electrostimulation added to pelvic floor muscle training can reduce leakage in Stress Urinary Incontinence (SUI)

DETAILED DESCRIPTION:
Among women with pelvic floor dysfunction, it has long been known that PFM training is the first-line therapy for stress incontinence. One of the difficulties that clinicians often find upon examination is that many women present a very weak pelvic floor and are unable to contract their PFM. There is overwhelming evidence to show that conservative treatment in the form of pelvic muscle exercises (and to a lesser degree, electrotherapy, and vaginal weight therapy) is effective in the treatment of stress urinary incontinence. To date, there is some evidence to support the use of electrical stimulation for stress urinary incontinence in women, but we are still very uncertain about the full potential of this treatment because of the low quality of the existing evidence.

ELIGIBILITY:
Inclusion Criteria:

* • Adult women (18 years old - 50 years old), with a Modified Oxford Score, determined by digital palpation, of 0 - 1, complaining leakage episode occurring more than once a week.

  * Between six and eighteen months after childbirth
  * Willing and able to be compliant with pelvic floor muscle exercise intervention (standard of care) for 12 weeks and to log compliance
  * Willing and able to undergo an extensive physical function evaluation

Exclusion Criteria:

* • pregnancy

  * severe neurological disease (Multiple Sclerosis, Parkinson's disease, spinal cord injury, major stroke or neuromuscular junction diseases)
  * previous operation for cancer or radiotherapy in the lower abdomen
  * Prior surgical intervention for urinary incontinence within the past 12 months
  * Hysterectomy within 12 months
  * voiding dysfunction
  * pelvic pain
  * severe prolapse (≥ grade 3)
  * recurrent urinary tract infection
  * pelvic or disseminated malignancies
  * women who were virgo intacta
  * women who declined vaginal examinations for any reasons
  * before four months of pregnancy
  * Having significant cognitive impairment or dementia
  * Unsafe to exercise (severe cardiopulmonary disease)
  * Unable/unwilling to provide informed consent
  * Patient has on physical examination, neurological and/or vaginal examination results which, in the opinion of the investigator, should exclude the subject.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Person's sense of self
Enrollment: 50 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Muscles (PFM) Strength | Baseline, four weeks, 6 and 12 months follow-up
  PFM strength by digital palpation done in the lithotomy position

SECONDARY OUTCOMES:
Frequency/volume chart | Baseline, four weeks, 6 and 12 months follow-up
  The change incontinence frequency (n.of episodes) deducted by frequency/volume chart
International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF) | Baseline, four weeks, 6 and 12 months follow-up
  Change of "International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF" scores, which varie from 0 (no impact of incontinence) to 19 (worst impact of incontinence in everyday life)

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Lamberti, MD, Principal Investigator — Azienda USL Piacenza
Locations (1):
- OSPEDALE FIORENZUOLA d'ARDA, Fiorenzuola d'Arda, PC, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data after deidentification

REFERENCES:
- [Result] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Result] Bo K. Pelvic floor muscle training is effective in treatment of female stress urinary incontinence, but how does it work? Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):76-84. doi: 10.1007/s00192-004-1125-0. Epub 2004 Jan 24. PMID 15014933